CLINICAL TRIAL: NCT00605605
Title: Anti-Inflammation & Vascular Endothelial Protection Effects of Dextromethorphan on Heavy Smoker
Brief Title: Vascular Endothelial Protection Effects of Dextromethorphan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Ping-Yen Liu/ Assitant Professor, National Cheng-Kung University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-93-28; 91-B-FA09-2-4 grant number
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2008-01-31 (Estimated); Status verified 2008-01

CONDITIONS: Atherosclerosis; Smoking; Inflammation
Keywords: endothelial function; atherosclerosis; smoking; inflammation; antioxidant
MeSH Terms: conditions — Atherosclerosis; Smoking; Inflammation | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — 120 mg/day, single once daily dose taken after breakfast by oral route
  Other Names: medicon for DM

SUMMARY:
To test the hypothesis that DM could have anti-inflammatory effect and thus achieve vascular protection effect on heavy smokers.

DETAILED DESCRIPTION:
Dextromethorphan (DM), an ingredient widely used in antitussive remedies, had been reported to reduce the inflammation-mediated degeneration of neurons. We recently found that DM can prevent vascular remodeling and neuron injury in animal models of carotid ligation and cerebral ischemia injuries, respectively. It was believed that its action was through the anti-oxidant and NADPH pathway to protect brain cells. However, the mechanism and actual effect on human vascular protection remained unclear.

To test the hypothesis that DM could have anti-inflammatory effect and thus achieve vascular protection effect on heavy smokers, this prospective study will be conducted to treat subjects with heavy smoking history with DM or not and evaluate the anti-inflammatory and the improvement of endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers who are currently smoking

Exclusion Criteria:

* personal history of hypertension or diabetes mellitus
* family history with
* documented premature cardiovascular events
* cardiovascular-associated sudden death
* total cholesterol > 240 mg/dL
* triglyceride > 200 mg/dL
* low-density lipoprotein > 160 mg/dL.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 1, 2, 3 and 6 month

SECONDARY OUTCOMES:
Surrogate end-points of the study: hs-CRP, sPLA2, matrix metalloproteinase-3, interleukin-6, tumor necrosis factor-alfa receptor II, GSH-Px, and urinary excretion of 8-PGF2alfa | 1, 2, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Yen Liu, MD, PhD, Principal Investigator — Assiatant Professor of National Cheng Kung University Medical Center
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan